CLINICAL TRIAL: NCT01828073
Title: Raltegravir Pharmacokinetics and Safety in Neonates
Brief Title: Evaluating the Safety and Pharmacokinetics of Raltegravir in Infants
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: P1097; 11790 (Registry Identifier: DAIDS ES); IMPAACT P1097
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Full term infants exposed in utero to maternal RAL: Infants, who were expected to be ≥2000 grams at birth (i.e. full-term) at time of enrollment, born to women with HIV-1 infection who received RAL 400 mg twice daily for at least two weeks prior to delivery and continued to receive ARVs during labor. The group also includes the mothers of these infants.
  Interventions: Drug: Raltegravir
- Cohort 2: LBW infants exposed in utero to maternal RAL: Infants, who were expected to be ≤2500 grams at birth (i.e. LBW) at time of enrollment, born to women with HIV-1 infection who received at least one dose of RAL 400 mg within 2 to 24 hours prior to delivery. The group also includes the mothers of these infants.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — No study-specific drugs were given to women or infants during this study. Women received RAL for clinical indications outside of the study.
  Other Names: RAL

SUMMARY:
The purpose of this study was to determine the washout pharmacokinetics (PK) and safety of in utero/intrapartum exposure to maternal raltegravir (RAL) in infants born to pregnant women with HIV infection who received RAL 400 mg twice daily. The study also provided data for the development of an infant RAL starting dosing regimen for IMPAACT P1110 (NCT01780831).

DETAILED DESCRIPTION:
Study participants were enrolled in two cohorts.

* Cohort 1 enrolled mother-infant pairs in which the infant was expected to be ≥2000 grams at birth (i.e. full term) at time of enrollment and the mother was living with HIV and received RAL 400 mg twice daily for at least 2 weeks prior to delivery and continued to receive antiretroviral (ARV) drugs during labor.
* Cohort 2 enrolled mother-infant pairs in which the infant was expected to be ≤2500 grams at birth [i.e. low birth weight (LBW)] at time of enrollment and the mother was living with HIV and received at least one dose of RAL 400 mg within 2 to 24 hours prior to delivery.

Cohorts 1 and 2 provided pharmacokinetics and safety data of in utero and intrapartum exposure to maternal RAL in full-term and LBW infants, respectively. Also, the study data were pooled with data from IMPAACT P1066 (NCT00485264) (Cohorts IV and V) and P1026s (NCT00042289) to determine the starting RAL dosing regimen for full-term and LBW infants in IMPAACT P1110 (NCT01780831).

The study initially opened accrual to Cohort 1 under protocol Version 1.0. Upon completion of accrual and follow-up of Cohort 1, the protocol was amended and accrual to and follow-up of Cohort 2 was under protocol Version 2.0.

No study-specific treatment was given to the participants during this study. The women (mothers) received RAL for clinical indications outside of the study. Infants received standard of care ARV therapy for prophylaxis of perinatal transmission of HIV as prescribed by their primary care physicians.

Cohort 1 mother-infant pairs were enrolled prior to delivery. The women were followed-up until discharge from the labor/delivery unit. Infants were followed from birth through 20 weeks after birth. If infant was eligible for PK sampling (see "Eligibility" section), blood samples were collected at 1-5, 8-14, 18-24, and 30-36 hours after birth. Protocol defined infant safety evaluations were at birth, and at 8-14 hours, 30-36 hours, 1 week and 20 weeks after birth.

Cohort 2 mother-infant pairs were enrolled prior to delivery or within 48 hours after delivery. The women were followed-up until discharge from the labor/delivery unit. Infants were followed from birth/entry through 6 weeks after birth. If infant was eligible for PK sampling, blood samples were collected at 1-6, 12-24, 36-48, 72-84, and 108-132 hours and 7-14 days after birth. Protocol defined infant safety evaluations were at entry/birth, and at 36-48 hours, 72-84 hours, 1 week and 6 weeks after birth.

For both cohorts, all infants regardless of whether they were eligible for PK sampling were included in the safety analyses. Infant safety data included adverse birth outcomes, signs/symptoms, diagnoses and chemistry/hematology test results. Protocol required chemistry tests were AST, ALT, serum creatinine, total bilirubin and direct bilirubin. Protocol required hematology tests were CBC with differential and platelet count. Also included in the safety data were additional laboratory events done outside of the study but considered by the site as relevant information.

For both cohorts, maternal blood and cord blood for RAL concentration testing were collected at delivery when specimen collection was possible. The optional genotypic testing (i.e. testing was done only if the mother consented) was limited to infants who were eligible for PK sampling. Information obtained about the effect of UGT1A1 polymorphisms on the PK of RAL was thought to provide a better understanding of the effect of genetics on the metabolism of RAL in neonates.

ELIGIBILITY:
Participant study inclusions and exclusion criteria are listed below.

Cohort 1 M-I pairs were enrolled prior to delivery so that only maternal study inclusion and exclusion criteria were assessed at enrollment.

Cohort 1: Maternal Study Inclusion Criteria

* Documentation of HIV-1 infection.
* Viable singleton pregnancy with gestational age of at least 35 weeks based on clinical or other obstetrical measurements with normal fetal anatomy
* Currently receiving RAL 400 mg twice daily for at least 2 weeks prior to enrollment in combination with other ARV agents for clinical care
* Plan to continue taking RAL in combination with other ARV agents through labor prior to delivery
* Willing and intends to deliver at the study-affiliated clinic or hospital
* Willing and able to sign informed consent for participation of herself and her infant. Participant must be of an age to provide legal informed consent as defined by the country in which she resides. If not, informed consent must be signed by a legal guardian.

Cohort 1: Maternal Study Exclusion Criteria

- Receipt of disallowed medications (phenobarbital, phenytoin, rifampin) within 4 weeks prior to enrollment

Cohort 1 Infants were enrolled prior to delivery so there were no infant study inclusion/exclusion criteria. However, only infants who met the following criteria were eligible for PK blood sampling. Infants ineligible for PK sampling remained in the study and were followed-up for safety.

Cohort 1: Infant PK Sampling Inclusion Criteria

* Infant born to women who received at least 2 weeks of RAL prior to delivery and continue to receive RAL during labor prior to delivery in addition to their other ARV drugs
* Infant birth weight of at least 2 kg
* Infant at least 37 weeks gestation at delivery
* Infant not receiving disallowed medications (phenobarbital, phenytoin, rifampin). If these medications are required for the infant's care, the infant will be ineligible for further PK sampling. PK samples will be obtained up to the time of the introduction of the disallowed medication.

Cohort 1: Infant PK Sampling Exclusion Criteria

- Infant has a severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the examining clinician

Cohort 2 enrolled M-I pairs at two time points: prior to delivery and within 48 hours after delivery.

* For M-I pairs enrolled prior to delivery, the maternal study eligibility criteria were assessed at enrollment. There were no infant study eligibility criteria. However, only infants who met the PK sampling eligibility criteria had PK blood sampling. Infants ineligible for PK sampling remained in the study and were followed-up for safety.
* For M-I pairs enrolled within 48 hours delivery, the maternal and infant study eligibility criteria were assessed at enrollment. A M-I pair was enrolled only if both the mother and the infant were eligible for the study. For multiple births, only infants who met the study eligibility criteria were enrolled.

Cohort 2: Maternal Study Inclusion Criteria: M-I pairs enrolled prior to delivery

* Documentation of HIV-1 infection.
* Viable singleton or multiple birth pregnancy based on clinical or other obstetrical measurements with infant birth weight anticipated to be less than or equal to 2,500 grams
* RAL is currently used as part of maternal ARV regimen and planned to continue through labor and delivery
* Willing and intends to deliver at the study-affiliated clinic or hospital
* Willing and able to sign informed consent for participation of herself and her infant. Participant must be of an age to provide legal informed consent as defined by the country in which she resides. If not, informed consent must be signed by a legal guardian.

Cohort 2: Maternal Study Exclusion Criteria: M-I pairs enrolled prior to delivery

- Receipt of disallowed medications (phenobarbital, phenytoin, rifampin) within 4 weeks prior to enrollment or intent to be on any of the disallowed medications prior to delivery.

Cohort 2: Infant PK Blood Sampling Eligibility Criteria: M-I pairs enrolled prior to delivery

Infants were enrolled prior to delivery so there were no infant study eligibility criteria. Only infants who met the following criteria were eligible for PK blood sampling:

* Infant born to woman who received at least one dose of RAL within 2 to 24 hours prior to delivery. Dose administered to mother must have been at least 2 hours prior to delivery to allow time for adequate absorption and distribution.
* Infant birth weight less than or equal to 2,500 grams
* Infant not receiving disallowed medications (phenobarbital, phenytoin, rifampin) as described in the protocol. If these medications are required for the infant's care, the infant will be ineligible for further PK sampling. PK data will be obtained up to the time of the introduction of the disallowed medication.
* Infant less than or equal to 48 hours of age
* Infant does not have any severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the examining clinician

Cohort 2: Maternal Study Inclusion Criteria: M-I pairs enrolled after delivery

* Documentation of HIV-1 infection.
* Received at least one dose of RAL within 2 to 24 hours prior to delivery
* Willing and able to sign informed consent for participation of herself and her infant. Participant must be of an age to provide legal informed consent as defined by the country in which she resides. If not, informed consent must be signed by a legal guardian.

Cohort 2: Maternal Study Exclusion Criteria: M-I pairs enrolled after delivery

- Receipt of disallowed medications (phenobarbital, phenytoin, rifampin) within 4 weeks prior to delivery

Cohort 2: Infant Study Inclusion Criteria: M-I pairs enrolled after delivery

* Infant birth weight less than or equal to 2,500 grams
* Infant less than or equal to 48 hours of age

Cohort 2: Infant Study Exclusion Criteria: M-I pairs enrolled after delivery

* Received disallowed medications (phenobarbital, phenytoin, rifampin)
* Infant has a severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the examining clinician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were enrolled in two cohorts.
  Cohort 1 enrolled Mother-Infant (M-I) pairs prior to delivery. Infants expected to be full term (i.e. ≥2000 grams at birth) born to women with HIV-1 infection who received RAL 400 mg twice daily for at least two weeks prior to delivery and continued to receive ARVs during labor, and their mothers, were enrolled to Cohort 1.
  Cohort 2 enrolled M-I pairs prior to delivery or within 48 hours after delivery. Infants expected to be LBW (i.e. ≤2500 grams at birth) born to women with HIV-1 infection who received at least one dose of RAL 400 mg within 2 to 24 hours prior to delivery, and their mothers, were enrolled to Cohort 2.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05-19; Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana F. Clarke, PharmD, Study Chair — Boston Medical Center
Locations (19):
- United States (12):
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Brazil (4):
  - Hospital Nossa Senhora da Conceicao NICHD CRS, Porto Alegre, Rio Grande do Sul
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- Soweto IMPAACT CRS, Johannesburg, Gauteng, South Africa
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai, Thailand

REFERENCES:
- [Background] Iwamoto M, Wenning LA, Petry AS, Laethem M, De Smet M, Kost JT, Merschman SA, Strohmaier KM, Ramael S, Lasseter KC, Stone JA, Gottesdiener KM, Wagner JA. Safety, tolerability, and pharmacokinetics of raltegravir after single and multiple doses in healthy subjects. Clin Pharmacol Ther. 2008 Feb;83(2):293-9. doi: 10.1038/sj.clpt.6100281. Epub 2007 Aug 22. PMID 17713476
- [Background] Wenning LA, Petry AS, Kost JT, Jin B, Breidinger SA, DeLepeleire I, Carlini EJ, Young S, Rushmore T, Wagner F, Lunde NM, Bieberdorf F, Greenberg H, Stone JA, Wagner JA, Iwamoto M. Pharmacokinetics of raltegravir in individuals with UGT1A1 polymorphisms. Clin Pharmacol Ther. 2009 Jun;85(6):623-7. doi: 10.1038/clpt.2009.12. Epub 2009 Mar 11. PMID 19279563
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, dated December 2004, Clarification August 2009 — https://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 participants were enrolled from 11 sites in the USA. Enrollment period was from May 2011 through September 2012.
  Cohort 2 participants were enrolled from 4 sites in Brazil, 1 site in South Africa, 1 site in Tanzania, 1 site in Thailand, and 3 sites in the USA. Enrollment period was from January 2015 through March 2018.
Groups:
- Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL: Infants, who were expected to be ≥2000 grams at birth (i.e. full-term), born to women with HIV-1 infection who received RAL 400 mg twice daily for at least two weeks prior to delivery and continued to receive ARVs during labor.
  Raltegravir: No study-specific drugs was given to women or infants during this study. Women received RAL for clinical indications outside of the study.
- Cohort 2: LBW Infants Exposed in Utero to Maternal RAL: Infants, who were expected to be ≤2500 grams at birth (i.e. LBW), born to women with HIV-1 infection who received at least one dose of RAL 400 mg within 2 to 24 hours prior to delivery.
  Raltegravir: No study-specific drugs were given to women or infants during this study. Women received RAL for clinical indications outside of the study.
Period: Overall Study
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Started | 22 | 18
Completed | 21 | 16
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: All infants
Groups:
- Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL: Infants, who were expected to be ≥2000 grams at birth (i.e. full-term), born to women with HIV-1 infection who received RAL 400 mg twice daily for at least two weeks prior to delivery and continued to receive ARVs during labor.
  Raltegravir: No study-specific drugs were given to women or infants during this study. Women received RAL for clinical indications outside of the study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 18 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  Enrolled prior to birth | 22 | 0 | 22
  Enrolled after birth | 0 | 18 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 13 | 9 | 22
  Unknown or Not Reported | 1 | 0 | 1
Birth Weight (g) [Count of Participants; unit: Participants]
  1500 - <2000 g | 0 | 7 | 7
  2000 - 2500 g | 1 | 11 | 12
  >2500 g | 21 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: PK Parameter: Neonatal RAL Elimination Half-life (T1/2)
Description: Time required for neonatal plasma concentration to decrease by one-half. T1/2 was estimated using the terminal 3 concentration-time points for each infant when available.
Time Frame: Infant blood specimens were collected at 1-5, 8-14, 18-24, and 30-36 hours after birth for Cohort 1; and at 1-6, 12-24, 36-48, 72-84, and 108-132 hours after birth, and on day 7-14 for Cohort 2.
Population: Infants with RAL concentration (conc) for whom T1/2 could be calculated. Excluded (i) 5 Cohort 1 infants: 2 had no data, 3 had data but could not calculate T1/2 (terminal RAL conc below level of quantification (BLQ), higher RAL conc at later collection time); and (ii) 1 Cohort 2 infants:1 had terminal RAL conc BLQ.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 17 | 17
Hours | 26.6 [9.3 to 184] | 24.4 [10.1 to 83]

2. Primary Outcome: Ratio of Cord Blood to Maternal Blood RAL Concentrations
Description: Ratio of the neonatal cord blood RAL concentration to the mother's plasma RAL concentration at birth
Time Frame: Maternal blood samples were scheduled to be collected within 1 hour after delivery and cord blood sample were collected immediately after cord was clamped
Population: Mother-Infant (M-I) pairs with maternal blood and cord blood samples. Excluded were (i) 3 Cohort 1 M-I pairs with neither cord blood nor maternal blood samples; and (ii) 16 Cohort 2 M-I pairs: 5 had neither cord blood nor maternal blood specimens, 11 had no cord blood specimen.
Measure: Median (Full Range); unit: ratio
Groups:
- Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL: Infants, who were expected to be ≥2000 grams at birth (i.e. full-term), born to women with HIV-1 infection who received RAL 400 mg twice daily for at least two weeks prior to delivery and continued to receive ARVs during labor. The group also includes the mothers of these infants.
  Raltegravir: No study-specific drugs were given to women or infants during this study. Women received RAL for clinical indications outside of the study.
- Cohort 2: LBW Infants Exposed in Utero to Maternal RAL: Infants, who were expected to be ≤2500 grams at birth (i.e. LBW), born to women with HIV-1 infection who received at least one dose of RAL 400 mg within 2 to 24 hours prior to delivery. The group also includes the mothers of these infants.
  Raltegravir: No study-specific drugs were given to women or infants during this study. Women received RAL for clinical indications outside of the study.
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 19 | 2
ratio | 1.48 [0.32 to 4.33] | 2.62 [1.04 to 4.20]

3. Primary Outcome: Number of Infants Who Met Composite Safety Endpoint (Grade 3/4 Adverse Event, Adverse Birth Outcome, Death)
Description: An infant was said to have met the composite safety endpoint if any of the following was observed:
  * adverse events (AEs) of Grade 3 or 4 as defined in DAIDS AE Grading Table
  * adverse birth outcomes including stillbirth and low birth weight (LBW), or
  * death.
  Stillbirth could only be observed on infants enrolled prior to delivery. Cohort 2 enrolled LBW infants and prematurity and growth restriction which were highly linked to LBW were considered as baseline events and not AEs or adverse birth outcome for Cohort 2 infants.
Time Frame: Assessed at entry through Week 20 for Cohort 1 infants and through Week 6 for Cohort 2 infants.
Population: All infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 22 | 18
Participants | 7 | 9
Statistical Analysis 1: Comparison: Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL; Point and 90% CI estimates of percentage of full term infants meeting the composite safety endpoint (grade 3/4 adverse event, adverse birth outcome, death); Test type: Other; Clopper-Pearson Confidence Interval (CI) = 31.82, 90% CI 2-sided [16.00 to 51.50] — With the small sample size, the CI estimate tend to be wide
Statistical Analysis 2: Comparison: Cohort 2: LBW Infants Exposed in Utero to Maternal RAL; Point and 90% CI estimates of percentage of full term infants meeting the composite safety endpoint (grade 3/4 adverse event, death); Test type: Other; Clopper-Pearson Confidence Interval (CI) = 50.00, 90% CI 2-sided [29.10 to 70.90] — With the small sample size, the CI estimate tend to be wide

4. Primary Outcome: Infant Total Bilirubin
Description: Total bilirubin measured from infant blood specimens.
Time Frame: Measured at 8-14 hours (Visit 1), 30-36 hours (Visit 2) and 1-2 weeks (Visit 3) after birth for Cohort 1; and at 36-48 hours (Visit 1), 72-84 hours (Visit 2) and 1 week (Visit 3)after birth for Cohort 2.
Population: Infants with total bilirubin results
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 22 | 18
mg/dL
  Visit 1: number analyzed (Participants) | 21 | 13
  Visit 1 | 3.7 [3.0 to 4.5] | 6.6 [5.9 to 8.1]
  Visit 2: number analyzed (Participants) | 19 | 13
  Visit 2 | 5.7 [3.8 to 7.0] | 10.7 [8.4 to 11.3]
  Visit 3: number analyzed (Participants) | 19 | 18
  Visit 3 | 2.7 [0.8 to 5.2] | 4.6 [2.2 to 9.3]

5. Primary Outcome: Infant Direct Bilirubin
Description: Direct bilirubin measured from infant blood specimens.
Time Frame: as for outcome 4
Population: Infants with Direct Bilirubin results
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 22 | 18
mg/dL
  Visit 1: number analyzed (Participants) | 18 | 16
  Visit 1 | 0.3 [0.2 to 0.4] | 0.5 [0.3 to 0.7]
  Visit 2: number analyzed (Participants) | 18 | 16
  Visit 2 | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.6]
  Visit 3: number analyzed (Participants) | 19 | 18
  Visit 3 | 0.3 [0.2 to 0.4] | 0.5 [0.4 to 0.6]

6. Primary Outcome: Number of Infants Who Received Treatment to Reduce Bilirubin or for Jaundice
Description: Assessment if infant received exchange transfusion, Phototherapy, or other treatment to reduce bilirubin or for jaundice
Time Frame: Assessed from entry through around week 1 after birth
Population: All infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
Number analyzed (Participants) | 22 | 18
Participants
  Exchange transfusion therapy | 0 | 0
  Phototherapy | 1 | 4
  Other treatment | 0 | 0

7. Secondary Outcome: Neonatal RAL Elimination (T1/2) by UGT1A1 Genotype Group (Normal VS Mutation)
Description: Neonatal RAL elimination was the time required for neonatal plasma concentration to decrease by one-half. Genotyping for polymorphisms of UGT1A1 were performed on infants who were eligible for PK sampling and were consented by their mothers/guardians(i.e. genotyping was optional) . The goal of the genotypic analysis is to determine if certain polymorphisms, particularly those with the UGT1A1*28/*28 genotype have slower RAL elimination than those with the UGT1A1*1/*1 genotype.
Time Frame: Genotype was assessed close to birth and if this is not possible at 1-2 wks after birth. PK samples were collected at 1-5, 8-14, 18-24 and 30-36 hrs after birth for Cohort 1; 1-6, 12-24, 36-48, 72-84 and 108-132 hrs after birth, and day 7-14 for Cohort 2.
Population: Infants with data on UGT1A1 genotype and RAL half-life (T1/2)
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Cohort 1 Infants With UGT1A1 Mutation: Cohort 1 (full term) infants with the presence of UGT1A1 *28/*28 genetic variant
- Cohort 1 Infants With Normal UGT1A1 Phenotype: Cohort 1 (full term) infants with the absence of UGT1A1 *28/*28 genetic variant
- Cohort 2 Infants With UGT1A1 Mutation: Cohort 2 (LBW) infants with the presence of UGT1A1 *28/*28 genetic variant
- Cohort 2 Infants With Normal UGT1A1 Phenotype: Cohort 2 (LBW) infants with the absence of the UGT1A1 *28/*28 genetic variant
Arm/Group | Cohort 1 Infants With UGT1A1 Mutation | Cohort 1 Infants With Normal UGT1A1 Phenotype | Cohort 2 Infants With UGT1A1 Mutation | Cohort 2 Infants With Normal UGT1A1 Phenotype
Number analyzed (Participants) | 8 | 6 | 9 | 7
Hours | 40.85 [13.55 to 82.05] | 32.75 [23.90 to 69.20] | 21.1 [18.4 to 26.3] | 39.7 [11.5 to 51.5]
Statistical Analysis 1: Comparison: Cohort 1 Infants With UGT1A1 Mutation vs Cohort 1 Infants With Normal UGT1A1 Phenotype; To investigate the relationship between neonatal RAL elimination and UGT1A1 genotype in full term infants; Test type: Other; p = 0.747, Wilcoxon (Mann-Whitney) — The study was not powered to do the comparison. This was an exploratory analysis
Statistical Analysis 2: Comparison: Cohort 2 Infants With UGT1A1 Mutation vs Cohort 2 Infants With Normal UGT1A1 Phenotype; To investigate the relationship between neonatal RAL elimination and UGT1A1 genotype in LBW infants; Test type: Other; p = 0.341, Wilcoxon (Mann-Whitney) — The study was not powered to do the comparison. This was an exploratory analysis

ADVERSE EVENTS:
Time Frame: Birth through 20 weeks and 6 weeks for Cohort 1 and Cohort 2, respectively.
Description: All Adverse Events (AEs) including diagnoses, signs/symptoms and abnormal laboratory test results mentioned in the "Study Description". LBW is an eligibility criterion for Cohort 2. Prematurity and growth restrictions, which were AEs linked with LBW, were defined in the protocol as baseline events for Cohort 2 infants and were excluded from the "Serious Adverse Events" and "Other Adverse Events tables" for Cohort 2.The DAIDS AE Grading Table (V1.0) and Expedited AE Manual (V2.0) were used.
Arm/Group | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 5/18
Other Adverse Events (participants affected / at risk) | 21/22 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL (N=22) | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL (N=18)
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 1
Hypospadias (Congenital, familial and genetic disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Infection prophylaxis (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Full Term Infants Exposed in Utero to Maternal RAL (N=22) | Cohort 2: LBW Infants Exposed in Utero to Maternal RAL (N=18)
Bradycardia neonatal (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 | 1
Congenital laryngeal stridor (Congenital, familial and genetic disorders) | 0 | 1
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 1 | 2
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Decreased activity (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 4
Bacterial sepsis (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 15 | 3
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatinine abnormal (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 5
Breath sounds abnormal (Investigations) | 2 | 0
Haemoglobin abnormal (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 8 | 5
Neutrophil count abnormal (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 5 | 6
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 6 | 4
Irritability (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2014-01-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT01828073/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT01828073/SAP_001.pdf